CLINICAL TRIAL: NCT02526823
Title: Clinical Application of Polyethylene Glycol Liposome Doxorubicin (PLD) in Primary Lymphoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Xin, Director of Department of Hematology, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShandongPH01
Record Dates: First submitted 2015-08-11; First posted 2015-08-18 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Lymphoma, Non-Hodgkin;Hodgkin Disease
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- R-CHOP/CHOPE or ABVD chemotherapy regimen (Active Comparator): R-CHOP/CHOPE every 21 days or ABVD every 28 days for total 6 courses
  Interventions: Drug: R-CHOP/CHOPE or ABVD chemotherapy regimen
- R-CDOP/CDOPE or DBVD chemotherapy regimen (Experimental): R-CDOP/CDOPE every 21 days or DBVD every 28 days for total 6 courses
  Interventions: Drug: R-CDOP/CDOPE or DBVD chemotherapy regimen

INTERVENTIONS:
Drug: R-CHOP/CHOPE or ABVD chemotherapy regimen — R-CHOP:
  Rituximab：375mg/m2，ivgtt，D0； Epirubicin：70 mg/m2，ivgtt，D1 ； Cyclophosphamide：750 mg/m2，ivgtt，D1； Vincristine: 1.4 mg/m2 ivgtt，D1 ； Prednison：100mg/d，po，D1-5；
  CHOPE:
  Epirubicin：70 mg/m2，ivgtt，D1 ； Cyclophosphamide：750 mg/m2，ivgtt，D1； Vincristine: 1.4 mg/m2 ivgtt，D1 ； Prednison：100mg/d，po，D1-5； Etoposide: 100 mg/（m2•d），ivgtt，D1-3;
  ABVD:
  Epirubicin：35 mg/m2，ivgtt，D1、15； Bleomycin：10 mg/m2，ivgtt，D1、15； Vincristine：1.4 mg/m2，ivgtt，D1、15； Dacarbazine：375mg/m2，ivgtt，D1、15；
  Arms: R-CHOP/CHOPE or ABVD chemotherapy regimen
Drug: R-CDOP/CDOPE or DBVD chemotherapy regimen — R-CDOP:
  Rituximab：375mg/m2，ivgtt，D0； PLD 30-40 mg/m2，ivgtt，D1 ； Cyclophosphamide：750 mg/m2，ivgtt，D1； Vincristine: 1.4 mg/m2 ivgtt，D1 ； Prednison：100mg/d，po，D1-5；
  CDOPE:
  PLD 30-40 mg/m2，ivgtt，D1； Cyclophosphamide：750 mg/m2，ivgtt，D1； Vincristine: 1.4 mg/m2 ivgtt，D1 ； Prednison：100mg/d，po，D1-5； Etoposide: 100 mg/（m2•d），ivgtt，D1-3;
  DBVD:
  PLD 15-20 mg/m2，ivgtt，D1； Bleomycin：10 mg/m2，ivgtt，D1、15； Vincristine：1.4 mg/m2，ivgtt，D1、15； Dacarbazine：375mg/m2，ivgtt，D1、15；
  Arms: R-CDOP/CDOPE or DBVD chemotherapy regimen

SUMMARY:
Anthracyclines were basic drugs in lymphoma treatment. However, their dose accumulation related cardiac toxicity limits their clinical application, especially adriamycin. Adriamycin has been gradually replaced by epirubicin. Polyethylene glycol liposome doxorubicin (PLD) can go into tumor tissues through tumor angiogenesis and produces targeted killing effect to tumor tissues. PLD has potential advantages in the treatment of malignant tumors,including lymphoma.

DETAILED DESCRIPTION:
Lymphoma is one of the most rapidly growing malignant tumors in the world. It was divided into two major categories (Hodgkin's lymphoma (HL) and non Hodgkin's lymphoma (NHL). Anthracyclines were basic drugs in lymphoma treatment. However, their dose accumulation related cardiac toxicity limits their clinical application, especially adriamycin. Adriamycin has been gradually replaced by epirubicin in malignant tumor treatment because of its similar effects and less toxic side effects. Polyethylene glycol liposome doxorubicin (PLD) is the liposome formulation of doxorubicin. Methoxy Polyethylene Glycol (MPEG) contained in liposome surface can decrease the peak plasma levels of free drugs, extend drugs circulation time in blood and reduce the chance of non-specific distribution to normal tissues. PLD goes into tumor tissues through tumor angiogenesis and produces targeted killing effect to tumor tissues. PLD has potential advantages in the treatment of malignant tumors. In lymphoma patients' therapy, the clinical application of PLD is expected to be a new method. Therefore, the investigators designed the randomized controlled clinical study and aimed to compare the efficacy and safety between PLD and epirubicin in primary B-NHL, peripheral T-cell lymphoma (PTCL) and HL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Primary B-NHL, PTCL (ALK+ anaplastic large cell lymphoma and NK(natural killer cell )/T cell lymphoma were excluded) or HL patients confirmed by histopathology;
2. Ages ≥18 years old, < 80 years old;
3. ECOG (Eastern Cooperative Oncology Group）score: 0-2
4. At least one measurable lesion;
5. Expected survival time≥3 months;
6. Liver function: transaminase≤2.5× upper limit of normal value，bilirubin≤1.5×upper limit of normal value;
7. Renal function: serum creatinine is 44-133 mmol/L;
8. Routine blood test：WBC≥3.0×109/L，Neutrophils≥1.5×109/L，Hb≥100g/L，Platelet≥80×109/L； LVEF≥50%;
9. New York Heart Association (NYHA) heart function classification is I-II grade
10. signed informed consent.

Exclusion Criteria:

1. Patients with severe complications or severe infection;
2. Invasion of central nervous system;
3. Patients with severe heart disease history, including ventricular tachycardia (VT), atrial fibrillation (AF), heart block, myocardial infarction (MI), congestive heart failure (CHF), coronary heart disease patients needed therapy;
4. patients with severe allergic constitution, or those who are allergic to or intolerant of drug composition in chemotherapy regimens; with other malignant tumors in the past 5 years;
5. patients received doxorubicin therapy, total cumulative dose of adriamycin was more than 300 mg/m2, total cumulative dose of epirubicin was more than 450 mg/m2;
6. Patients participate in other clinical studies;
7. Other patients who are not suitable for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with complete remission （CR） | After two 21-day or 28-day courses, up to 42 to 56 days.
  Sum of products of greatest diameters （SPD）was used to evaluate the therapy effect.Number of participants with CR was assessed by Cheson Standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology, Provincial Hospital Affiliated to Shandong University, Jinan, Shandong, China

REFERENCES:
- [Background] Lotrionte M, Biondi-Zoccai G, Abbate A, Lanzetta G, D'Ascenzo F, Malavasi V, Peruzzi M, Frati G, Palazzoni G. Review and meta-analysis of incidence and clinical predictors of anthracycline cardiotoxicity. Am J Cardiol. 2013 Dec 15;112(12):1980-4. doi: 10.1016/j.amjcard.2013.08.026. Epub 2013 Sep 25. PMID 24075281
- [Background] Italian Multicentre Breast Study with Epirubicin; Ambrosini G, Balli M, Garusi G, Demicheli R, Jirillo A, Bonciarelli G, Bruscagnin G, Fila G, Bumma C, Lacroix F, Buzzi F, Di Costanzo F, Padalino D, Brugia M, Calabresi F, Natali M, Cartei G, Chiesa G, Blasina B, Ciambellotti E, Moro G, D'Aquino S, Altavilla G, Adamo V, De Maria D, Falchi AM, Bertoncelli P, Farris A, Fiorentino M, Fornasiero A, Fosser V, Daniele O, Foggi CM, Speranza GB, Sartori S, Camilluzzi E, Gallo L, Poggio R, Secondo V, Gambi A, Grignani F, Capodicasa E, Lopez M, Papaldo P, Di Lauro L, Vici P, Marenco G, Folco U, Bonanni F, Marsilio P, Palazzotto G, Di Carlo A, Cusimano MP, Pastorino G, Puccetti C, Giusto M, Rausa L, Gebbia N, Palmeri S, D'Alessandro N, Saccani F, Becchi G, Schieppati G, Spinelli I, Tagliagambe A, Tonato M, Minotti V, Ardia A, Viaro D, De Micheli P, Zingali G, Sacchetti G, Intini C. Phase III randomized study of fluorouracil, epirubicin, and cyclophosphamide v fluorouracil, doxorubicin, and cyclophosphamide in advanced breast cancer: an Italian multicentre trial. J Clin Oncol. 1988 Jun;6(6):976-82. doi: 10.1200/JCO.1988.6.6.976. PMID 2897433
- [Background] Bai B, Huang HQ, Cai QQ, Wang XX, Cai QC, Lin ZX, Gao Y, Xia Y, Bu Q, Guo Y. Promising long-term outcome of gemcitabine, vinorelbine, liposomal doxorubicin (GVD) in 14-day schedule as salvage regimen for patients with previously heavily treated Hodgkin's lymphoma and aggressive non-Hodgkin's lymphoma. Med Oncol. 2013 Mar;30(1):350. doi: 10.1007/s12032-012-0350-5. Epub 2013 Jan 18. PMID 23329307
- [Background] Clozel T, Deau B, Benet C, Franchi P, Robin M, Madelaine I, Thieblemont C, de Kerviler E, Briere J, Brice P. Pegylated liposomal doxorubicin: an efficient treatment in patients with Hodgkin lymphoma relapsing after high dose therapy and stem cell transplation. Br J Haematol. 2013 Sep;162(6):846-8. doi: 10.1111/bjh.12428. Epub 2013 Jun 24. No abstract available. PMID 23789905
- [Background] Schmitt CJ, Dietrich S, Ho AD, Witzens-Harig M. Replacement of conventional doxorubicin by pegylated liposomal doxorubicin is a safe and effective alternative in the treatment of non-Hodgkin's lymphoma patients with cardiac risk factors. Ann Hematol. 2012 Mar;91(3):391-7. doi: 10.1007/s00277-011-1308-y. Epub 2011 Aug 18. PMID 21850390
- [Background] Fan Y, Lin NM, Luo LH, Fang L, Huang ZY, Yu HF, Wu FQ. Pharmacodynamic and pharmacokinetic study of pegylated liposomal doxorubicin combination (CCOP) chemotherapy in patients with peripheral T-cell lymphomas. Acta Pharmacol Sin. 2011 Mar;32(3):408-14. doi: 10.1038/aps.2010.217. PMID 21372831
- [Background] Rafiyath SM, Rasul M, Lee B, Wei G, Lamba G, Liu D. Comparison of safety and toxicity of liposomal doxorubicin vs. conventional anthracyclines: a meta-analysis. Exp Hematol Oncol. 2012 Apr 23;1(1):10. doi: 10.1186/2162-3619-1-10. PMID 23210520